CLINICAL TRIAL: NCT04307758
Title: Comparison of Strength Measurement in Intrinsic Foot Muscles With Break and Make Tests Using a Hand-held Dynamometer in Healthy Young Subjects
Brief Title: Strength Measurement in Intrinsic Foot Muscles With Break and Make Tests
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gokhan Yazici, Principal Investigator, Gazi University
Other Study IDs: GaziUni
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Adults
Keywords: Make and Break Test; Strength assessment; Hand held dynamometer; Intrinsic foot muscles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: Healthy subjects aged 18-35 years were enrolled in this study. The muscle strength assessment of the foot intrinsic muscles was assessed with the make test and the break test. The tests were performed with the hip and knee semiflexed in prone position with a hand-held dynamometer. The experimental protocols and methods were explained in detail to all subjects. All participants provided written informed consent in keeping with the ethical principles of the Declaration of Helsinki.
  Interventions: Other: Muscle Strength Assesment-Make Test; Other: Muscle Strength Assesment-Break Test

INTERVENTIONS:
Other: Muscle Strength Assesment-Make Test — For the make test, the examiner applies resistance in a fixed position and the person being tested exerts a maximum effort against the dynamometer and examiner. The examiner is only required to sustain an isometric contraction and read the highest value on an Hand Held Dynamometer.
  Other Names: Make Test
Other: Muscle Strength Assesment-Break Test — For the break test, the examiner applies resistance sufficient to overcome the maximum effort of the person being tested and cause the subject's joint to move in the opposite direction, which results in an eccentric contraction. During this test the limb must move at a constant velocity while the person being tested is asked to achieve a maximum contraction. In addition, the examiner must read the force output reading at the exact time the subject's limb begins to move from the Hand Held Dynamometer.
  Other Names: Break Test

SUMMARY:
The human foot is a complex structure, which serves functions such as support and mobility. These functions are accomplished through the deformation of the arch, which is controlled by intrinsic and extrinsic foot muscles. The intrinsic muscles have an important role in dynamic stabilization of the foot due to their structurally short force levers and small diameters. There are many studies reporting that foot intrinsic muscle weakness is directly related to pathologies such as structural or functional toe deformities, pes planus, hallux valgus, plantar fasciitis .Therefore it is essential to evaluate the strength of these muscles in an objective and reliable way.

DETAILED DESCRIPTION:
Two different methods are used in measuring muscle strength via a Hand Held Dynamometer; the "break test" and the "make test" . During these tests, the examiner and subject play opposite roles. During the make test, the subject applies maximal force against the examiner and the position is maintained by the examiner. During the break test, the subject holds the position of the muscle being evaluated and the examiner pushes until the subject's maximal force is overcome. In the two tests, force is applied differently; the dynamometer receives different amounts of force, and different results may be generated. Therefore, the aim of this study was to compare the reliability of intrinsic foot muscle strength assessment with break and make test in healthy young subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals,
* Category 1 and 2 according to the International Physical Activity Questionnaire
* Body mass index between the ranges ≥18.5 - <24.9

Exclusion Criteria:

* Any orthopedic or neurological disorder
* Previous history of lower extremity surgery
* Having low back pain
* Having vestibular or visual system problems
* Having hallux rigidus or limitus, having a hallux valgus angle over 15 degrees

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sedantary healthy individuals who do not have any orthopedic/neurologic lower extremity problems.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Foot intrinsic muscle strength with the make test | Once a day for two days.
  Reliability of the Make Test
Foot intrinsic muscle strength with the break test | Once a day for two days.
  Reliability of the Break test

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Yazici, Pt. PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No